CLINICAL TRIAL: NCT05178329
Title: Lifting Effect on Recovery After Mastectomy
Acronym: MUSKELI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anselm Tamminen (Other Government)
Responsible Party: Sponsor-Investigator, Anselm Tamminen, Consultant General Surgeon, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 93 /1801/2021
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-12

CONDITIONS: Seroma Complicating A Procedure
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The patients undergoing intervention exercise.
  Interventions: Behavioral: Lifting exercise
- Control Group (Placebo Comparator): The patients undergoing the normal exercise program
  Interventions: Behavioral: Standard exercise

INTERVENTIONS:
Behavioral: Lifting exercise — Patients are instructed for a light lifting exercise after mastectomy.
  Arms: Intervention group
Behavioral: Standard exercise — Standard exercise program after mastectomy
  Arms: Control Group

SUMMARY:
Breast cancer surgery has evolved towards ever more breast conserving direction. Even thought the surgical regime has become easier for the patient, many instructions given to the patient after the operation base on instructions, which have been used when the performed operations have been more burdensome.

Previously the patients have been instructed to lift only light objects after the operation, but according to the current knowledge, this instruction might be unnecessary.

The meaning of this study is to compare two patient groups to each other. The other group is instructed to avoid lifting, and the other group is given instructions to lift light weights several times daily.

In the study we compare will this have an effect on

1. incidence of upper limb lymphedema
2. seroma formation after surgery
3. quality of patients life after the surgery

Inclusion criteria is patients underoing mastectomy but no axillary clearance on day-care basis. Patietns will be randomized in two groups, the other as an intervention group and other as an control group. The patients are asked to fill a questionnaire considering recovery from the operation and possible wound healing problems. The amount of seroma is recorded. The volume of upper limbs is measured before and after the surgery.

The study is started in January 2022 and finished in December 2024.

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer diagnosis requiring mastectomy
* patients being operated in day-care regime

Exclusion Criteria:

* patients not eligible for day-care mastectomy
* patients undergoing axillary clearance operation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Volume of seroma formation after mastectomy. | 30 days

SECONDARY OUTCOMES:
Number of wound problems requiring intervention. | six months
Rate of lymphedema | one year
  Difference in upper limb volume after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Koskivuo, MD, PhD, Principal Investigator — TYKS

IPD SHARING:
Plan to Share IPD: No